CLINICAL TRIAL: NCT00880295
Title: Endoscopic vs Open Carpal Tunnel Release: Comparison of Patient Satisfaction, Outcomes, and Complications
Brief Title: Patient Outcomes With Endoscopic Versus Open Carpal Tunnel Release
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 24457
Record Dates: First submitted 2009-04-10; First posted 2009-04-13 (Estimated); Last update posted 2017-11-24 (Actual); Status verified 2017-11

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- endoscopic surgery (Active Comparator)
  Interventions: Procedure: endoscopic carpal tunnel release
- open surgery (Active Comparator)
  Interventions: Procedure: open carpal tunnel release

INTERVENTIONS:
Procedure: endoscopic carpal tunnel release — endoscopic surgery, which is standard of care for carpal tunnel release
  Arms: endoscopic surgery
Procedure: open carpal tunnel release — open surgery, which is standard of care for carpal tunnel release
  Arms: open surgery

SUMMARY:
Although some surgeons prefer one technique rather than the other, both endoscopic and open carpal tunnel release procedures are accepted as standard of care surgeries to relieve carpal tunnel syndrome. The investigator's research is designed to evaluate the significant difference in patient satisfaction between endoscopically-released wrists and open-released wrists. The goal of the study is to compare the two techniques using the following criteria:

1. Primary outcome: patient satisfaction via surveys used in prior publications
2. Secondary outcome: length of time to return to work
3. Secondary outcome: clinical data for recovery from carpal tunnel syndrome including a thorough physical exam and EMG's
4. Secondary outcome: complication rates

ELIGIBILITY:
Inclusion Criteria:

1. Patients between the ages of 18 and 75
2. Documented clinical and electromyography (EMG) proven carpal tunnel syndrome

Exclusion Criteria:

1. Recurrent carpal tunnel syndrome
2. Inflammatory arthropathy
3. Peripheral neuropathy
4. Diabetes
5. < 18 or > 75 years old
6. Pregnant at the time of enrollment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2009-03-23 (Actual); Primary Completion 2016-07-26 (Actual); Study Completion 2016-07-26 (Actual)

PRIMARY OUTCOMES:
Primary outcome: patient satisfaction via surveys used in prior publications | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Nogan, B.S., Principal Investigator — Penn State College of Medicine, Penn State Milton S. Hershey Medical Center
Locations (1):
- Penn State College of Medicine, Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States